CLINICAL TRIAL: NCT00990015
Title: A Phase 1, Randomized, Double-Blind, Sponsor-Open, Placebo-Controlled, Single-Dose Escalation Trial Evaluating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of PF-04308515 in Healthy Volunteers
Brief Title: A Phase 1 Single-Dose Escalation Study of PF-04308515 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: B0861001
Record Dates: First submitted 2009-10-02; First posted 2009-10-06 (Estimated); Last update posted 2010-02-01 (Estimated); Status verified 2010-01

CONDITIONS: Healthy Volunteers
Keywords: Safety; tolerability; pharmacokinetics/pharmacodynamics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-04308515 (Experimental)
  Interventions: Drug: PF-04308515
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-04308515 — Oral solution/suspension 0.1 mg up to potentially 350 mg QD at a single dose.
  Arms: PF-04308515
Drug: Placebo — Placebo solution/suspension to match active drug QD at a single dose.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety, tolerability, pharmacokinetics (understanding how a drug is absorbed and moves through the body) and pharmacodynamics (understanding the effects of a drug on certain target sites of activity in the body).

ELIGIBILITY:
Inclusion Criteria:

* Healthy males between 18 and 55 years, inclusive
* Healthy females between 18 and 44 years, inclusive.
* Women need to be surgically sterile

Exclusion Criteria:

* Evidence or history of clinically significant disease
* Post-menopausal women
* History of intolerance or significant adverse effects with glucocorticoids

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2009-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety, tolerability and pharmacokinetics (PK) of single-rising doses of PF-04308515 | 1 day
To characterize the pharmacodynamic (PD) effects of PF-04308515 on biomarkers | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0861001&StudyName=A%20Phase%201%20Single-Dose%20Escalation%20Study%20of%20PF-04308515%20in%20Healthy%20Volunteers